CLINICAL TRIAL: NCT00649090
Title: A Phase 4, Open-Label Exemestane Adjuvant Safety Surveillance Program: Adjuvant Exemestane (Aromasin) Treatment Following Previous Treatment With Tamoxifen in Postmenopausal Women With Estrogen Sensitive Primary Breast Cancer (IES Inclusion Criteria)
Brief Title: A Study to Evaluate the Safety of Adjuvant Treatment With Exemestane Following Previous Treatment With Tamoxifen in Postmenopausal Women With Estrogen Sensitive Primary Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5991077
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exemestane group (Active Comparator)
  Interventions: Drug: exemestane

INTERVENTIONS:
Drug: exemestane — Exemestane 25 mg oral tablet once daily for a maximum of 3 years

SUMMARY:
The purpose of this study was to give access to postmenopausal women with estrogen sensitive primary breast cancer to exemestane for the adjuvant treatment of breast cancer after the use of tamoxifen and to collect all serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients
* Patients with early breast cancer after adequate loco-regional treatment and eventual adjuvant chemotherapy, treated with tamoxifen for 2-3 years OR treated with tamoxifen for 2-3 years and consecutive exemestane treatment, provided the total duration of endocrine treatment is less than 5 years
* Estrogen receptor positive breast cancer patients
* Patients who remain free from disease following treatment with tamoxifen

Exclusion Criteria:

* Patients taking other drugs for the adjuvant treatment of breast cancer
* Patients taking hormone replacement therapy
* Donation of blood or blood products for transfusion during the 30 days prior to initiation of treatment with study drug, at any time during the program or 30 days after completion of treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1549 (Actual)
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Assess for serious adverse events | Months 3, 6, 12, 18, 24, and 30; Follow-up visit 28 days posttreatment

SECONDARY OUTCOMES:
Safety Surveillance Program | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- Belgium (53):
  - Pfizer Investigational Site, Aalst
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Arlon
  - Pfizer Investigational Site, Baudour
  - Pfizer Investigational Site, Bonheiden
  - Pfizer Investigational Site, Bouge
  - Pfizer Investigational Site, Boussu
  - Pfizer Investigational Site, Braine-l'Alleud
  - Pfizer Investigational Site, Brasschaat
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Charleroi
  - Pfizer Investigational Site, Chênée
  - Pfizer Investigational Site, Chimay
  - Pfizer Investigational Site, Dendermonde
  - Pfizer Investigational Site, Duffel
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Eupen
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Gilly (Charleroi)
  - Pfizer Investigational Site, Gosselies
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Herstal
  - Pfizer Investigational Site, Hornu
  - Pfizer Investigational Site, Huy
  - Pfizer Investigational Site, Kortrijk
  - Pfizer Investigational Site, La Louvière
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Libramont
  - Pfizer Investigational Site, Lier
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Mechelen
  - Pfizer Investigational Site, Merksem
  - Pfizer Investigational Site, Mons
  - Pfizer Investigational Site, Montigny-le-Tilleul
  - Pfizer Investigational Site, Mouscron
  - Pfizer Investigational Site, Namur
  - Pfizer Investigational Site, Ottignies
  - Pfizer Investigational Site, Rocourt
  - Pfizer Investigational Site, Roeselare
  - Pfizer Investigational Site, Seraing
  - Pfizer Investigational Site, Sint-Niklaas
  - Pfizer Investigational Site, Soignies
  - Pfizer Investigational Site, Tongeren
  - Pfizer Investigational Site, Torhout
  - Pfizer Investigational Site, Tournai
  - Pfizer Investigational Site, Turnhout
  - Pfizer Investigational Site, Verviers
  - Pfizer Investigational Site, Waregem
  - Pfizer Investigational Site, Wilrijk
  - Pfizer Investigational Site, Yvoir

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991077&StudyName=A%20Study%20to%20Evaluate%20the%20Safety%20of%20Adjuvant%20Treatment%20with%20Exemestane%20Following%20Previous%20Treatment%20withTamoxifen%20in%20Postmenopausal%20Women%20wi